CLINICAL TRIAL: NCT05130918
Title: The Efficacy of a Suppository Based on Phenolmicin P3 and Bosexil in Control of Irritative Symptoms in Patients Undergoing Thulium Laser Enucleation of Prostate: a Single-center, Randomized, Controlled, Open Label, Phase III Study
Brief Title: Efficacy of Mictalase® After ThuLEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Carlo di Nancy Hospital (Other)
Collaborators: Lampugnani Farmaceutici S.p.A. (Nerviano, Milan, Italy) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mictalase
Record Dates: First submitted 2021-11-02; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: BPH With Urinary Obstruction With Other Lower Urinary Tract Symptoms
Keywords: benign prostatic hyperplasia; BPH; laser enucleation; ThuLEP; LUTS; urinary tract infections
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenolmicin P3 and Bosexil (Experimental): Group in which patients were administered Phenolmicin P3 and Bosexil suppositories twice a day for 5 days, then once a day for other 10 days after thulium laser enucleation of prostate was performed.
  Interventions: Device: Phenolmicin P3 and Bosexil suppository
- Controls (No Intervention): Group in which patients were not administered Phenolmicin P3 and Bosexil suppositories after thulium laser enucleation of prostate was performed.

INTERVENTIONS:
Device: Phenolmicin P3 and Bosexil suppository — The suppository we herein investigated includes different active principles, namely: Bosexil®, that is a vegetal extract derived from the resin of the Boswellia serrata, a plant native to India. It has already been published that the Boswellic acids contained show anti-inflammatory and antioxidant properties in a variety of inflammatory diseases whose physio-pathological pathways are shared with those of prostatitis; phenolmicin P3 is a polyphenolic extract derived from beehive propolis, that also demonstrated anti-inflammatory and antioxidant properties in preclinical reports. It has also been reported to have the ability to create a microenvironment hostile to the reproduction of pathogenic bacteria.
  Other Names: Mictalase
  Arms: Phenolmicin P3 and Bosexil

SUMMARY:
In this single-center, prospective, randomized, open label, phase-III study, patients with indication to Thulium Laser Enucleation of Prostate were enrolled. The report conformed to CONSORT 2010 guidelines. Eligible patients were 1:1 randomized. Randomization defined Group A: patients who were administered Phenolmicin P3 and Bosexil suppositories twice a day for 5 days, then once a day for other 10 days; Group B: patients who did not receive the suppositories ("controls"). Study endpoints were evaluated at 15 and 30 days postoperation. Primary endpoint included evaluation of effects of the suppository on irritative symptoms by administering International Prostate Symptom Score (IPSS) with Quality of Life (QoL) questionnaire. Secondary endpoint included evaluation of effects on urinary tract infections by performance of urinalysis with urine culture.

ELIGIBILITY:
Inclusion Criteria:

- Patients with symptomatic benign prostatic hyperplasia deemed eligible for thulium laser enucleation of prostate.

Exclusion Criteria:

* patients with history of prostatitis,
* patients with history of neurogenic detrusor overactivity (as determined after urodynamic observation),
* patients diagnosed with prostate cancer,
* patients who underwent previous surgeries of the lower urinary tract,
* patients with indwelling catheter,
* patients with history of nephrolithiasis,
* patients with known or suspected hypersensitivity to Phenolmicin P3 and/or Bosexil
* patients experiencing occurrence of severe intraoperative complications.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The trial is conducted on a population of males who underwent surgical intervention for benign prostatic hyperplasia.
Enrollment: 111 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
IPSS | 15 and 30 days post-operation
  evaluation of effects of the suppository on irritative symptoms as assessed by eventual reduction in International Prostate Symptom Score (IPSS).
  Specifically, % reduction in absolute value of IPSS will be compared between the groups.
QoL | 15 and 30 days post-operation
  evaluation of effects of the suppository on Quality of life as assessed by eventual reduction in Quality of Life score.
  Specifically, % reduction in absolute value of QoL will be compared between the groups.

SECONDARY OUTCOMES:
Urinary Infection | 15 and 30 days post-operation
  evaluation of effects of the suppository on occurrence of urinary infections after thulium laser enucleation of prostate as assessed by urine culture.
  Specifically, the rates of positive urine culture will be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Bove, MD, Principal Investigator — San Carlo di Nancy Hospital
Locations (1):
- San Carlo di Nancy Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
The analysis of the data obtained within the trial will be subject of scientific publication

REFERENCES:
- [Derived] Bertolo R, Cipriani C, Vittori M, Carilli M, Maiorino F, Iacovelli V, Ganini C, Antonucci M, Signoretti M, Petta F, Panei M, Bove P. The efficacy of a suppository based on Phenolmicin P3 and Bosexil (Mictalase(R)) in control of irritative symptoms in patients undergoing thulium laser enucleation of prostate: a single-center, randomized, controlled, open label, phase III study. BMC Urol. 2022 Feb 12;22(1):19. doi: 10.1186/s12894-022-00974-0. PMID 35151280